CLINICAL TRIAL: NCT00492089
Title: A Randomized Phase II Trial of Bevacizumab to Control Brain Radiation Damage
Brief Title: Bevacizumab in Reducing CNS Side Effects in Patients Who Have Undergone Radiation Therapy to the Brain for Primary Brain Tumor, Meningioma, or Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCI-2009-00256; NCI-2009-00256 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000553135; 2006-0890 (Other: M D Anderson Cancer Center); 7955 (Other: CTEP); P30CA016672 (NIH); N01CM62202 (NIH)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2013-04

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Meningioma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Central Nervous System Germ Cell Tumor; Adult Choroid Plexus Tumor; Adult Diffuse Astrocytoma; Adult Ependymoma; Adult Grade II Meningioma; Adult Grade III Meningioma; Adult Malignant Hemangiopericytoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Papillary Meningioma; Adult Pineocytoma; Malignant Neoplasm; Meningeal Melanocytoma; Radiation Toxicity; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Adult Brain Tumor; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Basal Cell Carcinoma of the Lip; Stage I Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage I Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage I Lymphoepithelioma of the Nasopharynx; Stage I Lymphoepithelioma of the Oropharynx; Stage I Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Salivary Gland Cancer; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Nasopharynx; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Basal Cell Carcinoma of the Lip; Stage III Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage III Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Astrocytoma; Ependymoma; Meningioma; Oligodendroglioma; Choroid Plexus Neoplasms; Hemangiopericytoma, Malignant; Glioma; Pinealoma; Neoplasms; Radiation Injuries; Brain Neoplasms; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Bevacizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bevacizumab; Procedure: magnetic resonance imaging; Procedure: quality-of-life assessment
- Arm II (Placebo Comparator): Patients receive placebo IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: placebo; Procedure: magnetic resonance imaging; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm I
Drug: placebo — Given IV
  Other Names: PLCB
  Arms: Arm II
Procedure: magnetic resonance imaging
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: quality-of-life assessment
  Other Names: quality of life assessment

SUMMARY:
Bevacizumab may reduce CNS side effects caused by radiation therapy. This randomized phase II trial is studying how well bevacizumab works in reducing CNS side effects in patients who have undergone radiation therapy to the brain for primary brain tumor, meningioma, or head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine to what extent bevacizumab can reduce active radiation toxicity to the CNS in patients who have undergone cranial irradiation for primary brain neoplasm, meningioma, or head and neck cancer.

SECONDARY OBJECTIVES:

I. Determine to what extent this drug can reduce dexamethasone dependence in these patients.

II. Determine to what extent this drug can improve neurologic function in these patients.

III. Determine to what extent this drug can improve quality of life of these patients.

OUTLINE: This is a randomized, placebo-controlled, crossover, double-blind study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Patients in arm II who have failed to respond to treatment at 6 or 12 weeks may cross over to arm I and receive 2 courses of bevacizumab as in arm I. Patients in arm I (including crossover patients) who have responded to treatment may receive 2 additional courses of bevacizumab.

Patients undergo MRI after courses 2 and 4.

Quality of life and neurologic function are assessed at baseline, periodically during study treatment, and at 12 and 24 weeks after completion of study treatment.

After completion of study treatment, patients are followed at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of bleeding diathesis or coagulopathy
* Fertile patients must use effective contraception during and for >= 2 months after completion of study therapy
* No diarrhea >= grade 1
* Histologically confirmed primary brain neoplasm, meningioma, or head and neck cancer [WHO grade 2 or 3 disease--no WHO grade 4 primary brain neoplasms (i.e., glioblastoma or gliosarcoma)]
* Patients with head and neck cancer must not have any of the following:

  * Evidence of metastatic disease
  * Evidence of tumor invasion to major vessels (e.g., the carotid)
  * History of bleeding related to tumor or radiotherapy during or after completion of radiotherapy
* Must have undergone cranial irradiation
* Must have radiographic evidence to support the diagnosis of radiation necrosis and/or surgical biopsy evidence of necrosis without tumor within the past 2 months
* Must have evidence of progressive neurologic signs or symptoms appropriate to the location of the radiation necrosis
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury within the past 28 days
* No evidence of active CNS hemorrhage
* Karnofsky performance status 60-100%
* No clinically significant cardiovascular disease, including any of the following:

  * Inadequately controlled hypertension (i.e., systolic BP > 140 mm Hg and/or diastolic BP > 90 mm Hg despite antihypertensive medication)
  * Large vessel cerebrovascular accident within the past 6 months
  * Myocardial infarction or unstable angina within the past 6 months
* No clinically significant cardiovascular disease, including any of the following:

  * NYHA class II-IV congestive heart failure
  * Serious or inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm or history of aortic dissection)
  * Clinically significant peripheral vascular disease
* At least 6 months since prior radiotherapy
* Platelet count > 75,000/mm^3
* Granulocyte count > 1,500/mm^3
* Creatinine < 1.0 times ULN
* AST < 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Prior chemotherapy for tumor allowed
* Prior tyrosine kinase inhibitors of VEGF receptor (VEGFR) allowed
* More than 28 days since prior and no concurrent major surgical procedure or open biopsy
* Concurrent dexamethasone allowed provided patient is on a stable dose for >= 1 week prior to study entry
* Concurrent full-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 allowed provided the following criteria are met:

  * In-range INR (usually between 2 and 3) and patient is on a stable dose of oral anticoagulant for 1 week or on a stable dose of low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding
* Concurrent full-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 allowed provided the following criteria are met: No evidence of serious or nonhealing wound, ulcer, or bone fracture
* No concurrent chemotherapy or tyrosine kinase inhibitors of VEGFR
* No prior bevacizumab
* More than 7 days since prior core biopsy
* History of seizures allowed provided the patient is receiving anticonvulsant therapy
* Hemoglobin >= 9.0 g/dL
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Loghin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 20, 2007 to December 07, 2009. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 15 patients enrolled, four participants were excluded from the study.
Groups:
- Arm A: Bevacizumab: Bevacizumab 7.5 mg/m^2 intravenous (IV) every 3 weeks.
- Crossover Arm B: Placebo First, Then Bevacizumab: Placebo IV every 3 weeks for two courses, crossover at 6 weeks to receive Bevacizumab 7.5 mg/m^2 IV as in Arm A.
Period: First Intervention (6 Weeks)
Arm/Group | Arm A: Bevacizumab | Crossover Arm B: Placebo First, Then Bevacizumab
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Arm A: Bevacizumab | Crossover Arm B: Placebo First, Then Bevacizumab
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Bevacizumab | Crossover Arm B: Placebo First, Then Bevacizumab | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Full Range); unit: years] | 43 [39 to 59] | 47 [39 to 70] | 47 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response ( > 25% Reduction in T2 Flair) From Baseline to Evaluation at 6 Weeks Post Treatment
Description: Change in magnetic resonance imaging (MRI) from baseline to evaluation at 6 weeks for participants where MRI changes are based on the size of edema (T2 FLAIR) and Gd-contrast enhancement (lesion diameter and perfusion/dynamic). A 25% reduction in T2 flair volume constitutes a response for study.
Time Frame: Baseline to 12 weeks
Population: Analysis was conducted per protocol. The participants in the Crossover Arm were evaluated after receiving the Bevacizumab treatment as described in the arm description.
Measure: Number; unit: participants
Groups:
- Crossover Arm B: Placebo Then Bevacizumab: Placebo IV every 3 weeks for two courses, crossover at 6 weeks to receive Bevacizumab 7.5 mg/m^2 IV as in Arm A
Arm/Group | Arm A: Bevacizumab | Crossover Arm B: Placebo Then Bevacizumab
Number analyzed (Participants) | 5 | 6
participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 2 years and 9 months
Groups:
- Bevacizumab: Bevacizumab 7.5 mg/m^2 intravenous (IV) every 3 weeks
- Placebo: First Intervention Placebo IV (only) every 3 weeks for two courses
Arm/Group | Bevacizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 4/11 | 0/6
Other Adverse Events (participants affected / at risk) | 5/11 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=11) | Placebo (N=6)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=11) | Placebo (N=6)
Hypertension (Cardiac disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Elevated alanine aminotransferase (ALT) (Hepatobiliary disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less